CLINICAL TRIAL: NCT00005009
Title: Evaluation of the Safety and Immunogenicity of Varivax® (Live-Attenuated Varicella-Zoster Virus Vaccine) in Pediatric Renal Transplant Recipients
Brief Title: Evaluation of the Safety of Varivax® in Pediatric Renal Transplant Recipients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Merck Sharp & Dohme LLC (Industry); Cooperative Clinical Trials in Pediatric Transplantation (Network); North American Pediatric Renal Trials and Collaborative Studies (NAPRTCS) (Unknown); NIAID Vaccine and Treatment Evaluation Units (VTEUs) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DAIT VZV
Record Dates: First submitted 2000-03-28; First posted 2001-08-31 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Kidney Transplant Recipients
Keywords: pediatric renal transplant recipients; varicella zoster virus (VZV) vaccine; herpes zoster vaccine; VZV susceptible; safety; immunogenicity
MeSH Terms: conditions — Chickenpox | interventions — Chickenpox Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Varivax® (Experimental): 0.5 mL of Varivax administered subcutaneously in the right upper arm (deltoid region).
  Interventions: Biological: Varivax®

INTERVENTIONS:
Biological: Varivax® — Each participant will receive 2 doses of Varivax 6 to 8 weeks apart.
  Other Names: live-attenuated varicella zoster virus vaccine; varicella zoster virus vaccine; Oka-Merck live virus vaccine

SUMMARY:
The purpose of this study is to find out whether Varivax is safe for use in children with kidney transplants and whether it protects children from serious infection. Varivax is a vaccine against varicella zoster virus (VZV), the virus that causes chickenpox (varicella) and shingles (zoster).

Healthy children are already receiving Varivax shots to protect them from chickenpox. Few children with kidney transplants have received Varivax because doctors have been concerned that Varivax might cause serious reactions in them. On the other hand, VZV infection can be a life-threatening disease in these children. For this reason, doctors ultimately want to learn whether Varivax might safely prevent VZV infections in children who have had kidney transplants.

DETAILED DESCRIPTION:
Pediatric renal transplant patients face a lifetime of immunosuppressive therapy that place them at high risk for potentially life-threatening infection by primary varicella zoster virus (VZV). Treatment for acute episodes of VZV infection is possible but expensive and provides no long-term protection. Furthermore, therapy to overcome VZV infections can lead to renal graft rejection.

Varivax has proven safe, immunogenic, and effective in the normal host and has been recommended for universal administration in the general population at age 12 months. It is not currently labeled for use in immunocompromised patients. However, recent studies in pediatric leukemia and pediatric renal transplant patients suggest that attenuated live vaccine can confer protection with minimal adverse events even in the presence of immunosuppression, providing encouragement for more careful studies of VZV immunization in renal transplant patients. This study aims to quantify the safety and immunogenicity of Varivax in the population of pediatric renal transplant patients least susceptible to VZV infection, i.e., those on minimal maintenance immunosuppression and at least 1 year out from transplant.

Patient enrollment is staged to allow study physicians to closely monitor patients for signs of disseminated varicella reactions or graft rejection. Initially only 1 patient will be enrolled in the study. If the first patient reaches Week 8 without a severe adverse reaction, 3 study centers will then enroll 3 additional patients. If 8 weeks later these 3 patients have had no severe adverse reactions, the same 3 study centers will enroll 3 more patients. At the end of this period, having ascertained the safety of the vaccine in the first 7 patients, the study will be opened to the remaining centers. Patients receive 2 doses of Varivax 6 to 8 weeks apart. Each week for 6 to 8 weeks after the first vaccine dose, the patient undergoes venipuncture and clinical assessment to characterize renal graft and liver function and identify any signs of varicella infection. Additional telephone follow-up occurs on Day 4 and twice weekly thereafter. Parents or guardians monitor the patient for evidence of rash or fever and immediately report any rashes or fevers to study physicians. If, after 6 to 8 weeks, the patient demonstrates no severe reactions to the vaccine and requires no antiviral therapy, the patient receives the second vaccine dose. The patient again receives weekly on-site and telephone follow-up for 6 weeks. Other visits occur 9 weeks and 14 weeks after the second vaccine dose and 1 year after the first vaccine dose. At these visits the patient undergoes venipuncture and clinical assessment to identify potential rejection events or varicella infection and to characterize VZV antibody responses and cytokine changes in response to the vaccine.

ELIGIBILITY:
Inclusion Criteria:

Your child may be eligible for this trial if he/she:

* Had a kidney transplant 1 year ago or more;
* Is between 2 and 21 years of age (parent or guardian's signed informed consent required if under 18);
* Is taking stable, maintenance doses of immunosuppressive drugs for his/her kidney transplant; and
* Is generally in good health.

Exclusion Criteria:

Your child will not be eligible for this trial if he/she:

* Has had any rejection episodes in the last 6 months or has other problems with their kidneys;
* Was in the hospital for a major infection in the last 30 days;
* Has a history of VZV infection, including chicken pox or shingles;
* Has ever received a VZV vaccine, including Varivax®;
* Lives with a person whose immune system does not work well;
* Is allergic to certain medications;
* Is unable to return for the prescribed follow-up check-ups;
* Has no phone or pager; or
* Has had blood or plasma transfusions or taken certain drugs in the last 6 months.

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 1998-02; Primary Completion 2001-06-16 (Actual); Study Completion 2001-06-16 (Actual)

PRIMARY OUTCOMES:
Immediate adverse reactions | 30 minutes post vaccination
Varicella related adverse reactions | 1 year
  1. Fever and local (<1 inch from inoculation site) lesions
  2. Fever and lesions outside the 1 inch inoculation site
  3. Lesions outside the 1 inch inoculation site
  4. Clinical signs of pneumonitis
  5. Clinical or chemical signs of hepatitis
  6. Development of thrombocytopenia
Rejection events | 1 year
  1. Increase in creatinine
  2. Renal biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Amir Tejani, MD, Study Chair — North American Pediatric Renal Transplantation Study (NAPRTCS); Beverly L. Connelly, MD, Study Chair — Vaccine and Treatment Evaluation Unit (VTEU)-Cincinnati Children's
Locations (4):
- United States (4):
  - University of Alabama at Birmingham - Vaccine and Treatment Evaluation Unit (VTEU), Birmingham, Alabama
  - Boston Children's Hospital - Vaccine and Treatment Evaluation Unit (VTEU), Boston, Massachusetts
  - University of Michigan - Vaccine and Treatment Evaluation Unit (VTEU), Ann Arbor, Michigan
  - University of Texas Health Science Center at San Antonio - Vaccine and Treatment Evaluation Unit (VTEU), San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Participant level data and additional relevant materials are available to the public in the Immunology Database and Analysis Portal (ImmPort). ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) website — https://www.niaid.nih.gov/about/dait
- See also: NIAID Vaccine and Treatment Evaluation Units (VTEUs) — https://www.niaid.nih.gov/networks-collaborations/vaccine-and-treatment-evaluation-units-vteus
- Available data/document: Individual Participant Data Set: SDY357 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY357 — ImmPort study identifier is SDY357.
- Available data/document: Study Protocol: SDY357 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY357 — ImmPort study identifier is SDY357
- Available data/document: Study summary, -design, -demographics, -lab tests, -study files: SDY357 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY357 — ImmPort study identifier is SDY357